CLINICAL TRIAL: NCT04951687
Title: The Acute and Chronic Effects of Ecologic Barrier© on Mood and Cognition
Brief Title: Acute and Chronic Effects of Ecologic Barrier© on Mood and Cognition
Acronym: ProCog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Winclove Probiotics B.V. (Industry)
Responsible Party: Principal Investigator, Prof Claire Williams, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2-2020
Record Dates: First submitted 2021-05-11; First posted 2021-07-07 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Change; Mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active: Ecologic Barrier© (Experimental): Dietary supplement: Ecologic Barrier©
  Ingredients: maize starch, maltodextrin, vegetable protein, potassium chloride, magnesium sulphate, manganese sulphate, and probiotic bacteria (B. bifidum W23, B. lactis W51, B. lactis W52, L. acidophilus W37, L. brevis W63, L. casei W56, L. salivarius W24, Lc. lactis W19, Lc. lactis W58).
  Subjects will consume 2g (5 billion CFU)/day of Ecologic Barrier©. The intervention is a powder which is sealed in sachets and an be stored at room temperature by participants. Subjects are to mix into warm water and drinking alongside a meal.
  Interventions: Dietary Supplement: Ecologic Barrier©
- Placebo (Placebo Comparator): Dietary supplement: placebo powder
  Ingredients: maize starch, maltodextrin, vegetable protein, potassium chloride, magnesium sulphate, manganese sulphate.
  As with the active treatment, the intervention is a powder which is sealed in sachets and an be stored at room temperature by participants. Subjects are to mix into warm water and drinking alongside a meal.
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Ecologic Barrier© — 5x10^9 CFU/ 2g per day of Ecologic Barrier©
  Arms: Active: Ecologic Barrier©
Dietary Supplement: Placebo powder — matched placebo
  Arms: Placebo

SUMMARY:
This study aims to investigate the acute and chronic effects of an 8 week probiotic intervention (Ecologic Barrier©) on mood and cognitive outcomes in healthy adults.

DETAILED DESCRIPTION:
This study will employ a double-blind, randomised, placebo-controlled crossover design to investigate the acute and chronic effects of an 8 week probiotic intervention (Ecologic Barrier©) on mood and cognitive outcomes in healthy older adults. A total of 30 participants will be enrolled and counterbalanced to receive the active probiotic treatment (2g per day Ecologic Barrier©) or a matched placebo in the first arm, before having a 4 week washout period and continuing with 8 weeks of the second treatment not consumed within the first arm. Outcome measures will be assessed at baseline, 24 hours and 8 weeks within each arm. These will include cognitive measures of affective processing, immediate and delayed verbal memory, visuospatial working memory and executive functions, and mood measures of depressive symptoms, cognitive reactivity, anxiety, stress and general mood. In addition, faecal samples will be collected at all timepoints in order to explore faecal microbiota profiles before and after probiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 65 - 80
* Agree not to not consume probiotic or prebiotic supplements or live yoghurt throughout the course of study.
* Proficient in the English language

Exclusion Criteria:

* Already a habitual user of probiotics
* Antibiotic treatment within last 3 months
* Current diagnosis of and not currently receiving treatment for mental health disorder
* Gastrointestinal disorder
* Allergic to any ingredient of the active or placebo treatment
* Regular smoker
* Diabetes mellitus

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Corsi Block Tapping Test performance | Baseline, 24 hours and 8 weeks
  A standardised assessment of visuospatial working memory. The task comprises nine identical squares fixed in a random arrangement on a screen. Participants observe sequences of between two and nine blocks, which they then reproduce as accurately as possible. The dependent variable is the number of blocks pointed out in the correct order. Four versions of each sequence length are presented during the task. A novel sequence will be presented on each occasion, the order of which will be counterbalanced across participants.
Change in Immediate Word Recall from the Rey Auditory Verbal Learning Task | Baseline, 24 hours and 8 weeks
  Participants will be presented with a sequential list of 15 words, at a rate of 1 word per second. The participant will then have 60s to say out loud as many of these words as possible, with the resulting score recorded as a percentage of accuracy.

SECONDARY OUTCOMES:
Rey Auditory Verbal Learning Task - Delayed Word Recall | Baseline, 24 hours and 8 weeks
  After a period of time subject are asked to recall as many words as possible from list A
Rey Auditory Verbal Learning Task - Word Recognition | Baseline, 24 hours and 8 weeks
  Following the delayed word recall, words from list A, list B and novel words are displayed sequentially on the screen and participants are asked to indicate which words were from list A only.
Switching task | Baseline, 24 hours and 8 weeks
  This task requires executive function and sustained attention, and provides a measure of cognitive flexibility. Participants view a circle with 8 equally spaced radii 2 of which form a bold bisecting line. Numbers are chosen randomly from a set of 1-4 & 6-9 and displayed sequentially in a clockwise direction. A response of higher or lower than 5 is made for trials below the bold line, and even or odd for numbers above the line. Outcome measures include overall accuracy and reaction time (RT) on correct trials, as well as accuracy and RT on trials where there is a 'switch cost' from stimuli moving from below to above the bold line and vice versa.
Go/No Go task | Baseline, 24 hours and 8 weeks
  This task measures executive function - specifically the ability to inhibit or withhold a response to no-go stimuli. Both a neutral block (white circles) and an emotional block (happy and fearful faces from the FACES database) are included here, in order to explore any additional influence of emotional stimuli on inhibitory responses. Outcome measures include accuracy and reaction time (RT). Accuracy and reaction times in the emotional blocks may also be correlated with responses to mood measures.
Leiden Index of Depression Sensitivity revised (LEIDS-r) | Baseline, 24 hours and 8 weeks
  A validated questionnaire measure of cognitive reactivity. The LEIDS-r comprises of 34 items which the participant rate on a scale from 0-4 to indicate how strongly each statement applied to them when they are feeling somewhat sad.
Positive and Negative Affect Schedule expanded (PANAS-x) | Baseline, 24 hours and 8 weeks
  A validated self-report measure of affective state. The PANAS comprises of two distinct affective states (positive and negative), as well as 11 individual affective states (fear, guilt, sadness, surprise, hostility, shyness, joviality, self-assurance, attentiveness, fatigue and serenity. Subjects use a likert scale from 1 - 5 to indicate how the word relates to how they are currently feeling. As this analysis is exploratory all affective states will be explored.
State Trait Anxiety Inventory | Baseline, 24 hours and 8 weeks
  A well validated scale for assessing self-reported state and trait anxiety. In line with the study objectives, only the state items will be used to assess current feelings of anxiety in the participants. This includes 10 items which are rated using a 4-point likert scale.
Perceived Stress Scale | Baseline and 8 weeks
  A validated 10 item scale for self-reporting levels of perceived stress over the last month. Items are rated using a 5-point likert scale.
Centre for Epidemiological Studies Depression Scale (CESD) | Baseline and 8 weeks
  A validated, brief self report measure of depressive symptoms commonly used to assess sub-clinical levels of low mood. Items are responded to using a 4-point likert scale. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.

OTHER OUTCOMES:
Faecal sample analysis | Baseline, 8 weeks
  16S rRNA sequencing for classification and quantification of faecal bacteria
Montreal Cognitive Assessment | Baseline (arm 1 only)
  The Montreal Cognitive Assessment (MoCA) is a short cognitive screening tool to indicate current cognitive status. It is similar to the Mini Mental State Examination, but more sensitive to Mild Cognitive Impairment. Results will not be used to screen for eligibility, but baseline MoCA score may be included as covariate.
Epic-Norfolk Food Frequency Questionnaire (FFQ) | Baseline (arm 1 only)
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK, which is particularly important to explore in order to understand how the probiotic supplement may interact with diet and gut microbiome diversity. Data will be processed using the FETA software.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lamport, Associate Prof, Principal Investigator — University of Reading; Saskia Van Hemert, Study Director — Winclove Probiotics B.V.
Locations (1):
- School of Psychology and Clinical Languages, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eastwood J, van Hemert S, Stolaki M, Williams C, Walton G, Lamport D. Exploring the acute and chronic effects of a multistrain probiotic supplement on cognitive function and mood in healthy older adults: a randomized controlled trial. Am J Clin Nutr. 2025 Jun;121(6):1268-1280. doi: 10.1016/j.ajcnut.2025.04.002. Epub 2025 Apr 11. PMID 40222448

DOCUMENTS (1):
  • Study Protocol (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04951687/Prot_000.pdf